CLINICAL TRIAL: NCT04967729
Title: The Utility of Self-administered Lung Ultrasound in Patients With COVID-19
Brief Title: COVID-19 and Lung Ultrasound Utility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rocket Doctor Inc. (Other)
Responsible Party: Principal Investigator, William Cherniak, Principal Investigator, Rocket Doctor Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-2711-6322-3
Record Dates: First submitted 2021-07-07; First posted 2021-07-20 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- LUS ultrasound and standard of care (Other): Subjects will perform a lung ultrasound in order to determine the ability of patients to take an ultrasound from their homes. The lung ultrasound will be coupled with telehealth clinical support to monitor the severity of COVID-19 patients and provide standard of care. All subjects will receive the lung ultrasound technology and daily calls for teleguidance through the ultrasound and standard of care to monitor symptoms.
  Interventions: Device: Device: Butterfly iQ

INTERVENTIONS:
Device: Device: Butterfly iQ — The Butterfly iQ is an ultrasound system that enable diagnostic ultrasound imaging and measurement of anatomical structures and fluids of adult and pediatric patients. It is a non-invasive device and does not impose any health hazards.

SUMMARY:
Ultrasounds are usually done by a specially trained health professional in the hospital or emergency department (ED) setting. Using a novel single-probe device, the ultrasound can be plugged into an iOS / Android device. The purpose of this research is to assess the usefulness of lung ultrasound imaging, performed by the patient in the home setting for the management of the COVID-19 disease using this novel highly-portable ultrasound.

DETAILED DESCRIPTION:
This will be a prospective self-controlled design. The study subjects will receive a telehealth visit from a healthcare provider (HCP) to assess for any change in their COVID-19 symptoms. The HCP will recommend the patient remain at home, or to go to an emergency department based on standard of care and clinical decision making. Subsequently, the study subjects will receive a teleguidance session with a Radiologist who is trained in lung ultrasound (LUS) in order to obtain images of their chest. The physician performing LUS remotely will report LUS findings in a standard quality assurance (QA) document, including image quality, interpretation, and recommendations. This QA report will be study data and not shared with the patient. The two providers will be blinded, except when there is a disagreement between the Telemed LUS and clinical interview.

The study staff will determine when this disagreement occurs. They will notify the study investigators and radiologist, who will then discuss and come to an agreement within 24 hours. If deemed concerning, they will then contact the HCP and unblind them as to the radiographic findings. There will be no delay in medical care advised by the subject's HCP.

Specifically, the nurse will inform the HCP by a phone call that the physician performing LUS remotely found a significant change in LUS findings. The HCP will then be given access to the LUS report (as well as images if desired), and will review the decision to seek medical care with the telemed doctor.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older and able to provide a valid informed consent.
* Must have a nasal swab positive RT-PCR for COVID-19
* Must have access to Wi-Fi at home

Exclusion Criteria:

* Subjects unwilling or unable to directly provide consent.
* The following vulnerable study subject populations will not be eligible: prisoners, mentally impaired, or disadvantaged groups.
* Any condition deemed by the principal investigator, in his or her judgment, that may impact the subject's ability to meet the requirements necessary to collect the exam data required.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
The efficacy of image-acquisition for patient-performed lung ultrasound as assessed by a standard Quality Assurance, including image quality, interpretation, and recommendations. | 14 days
  Patients will perform a lung ultrasound with teleguidance from a medical professional. This will be taken daily and monitored by an expert clinician who can guide based on the remote live transmission and probe position. The efficacy of the images obtained will be assessed using a standard Quality Assurance report using Soldati scoring which will be completed and synthesized following each appointment during the fourteen day period.

SECONDARY OUTCOMES:
Correlate LUS radiographic findings with patient outcomes. | 14 days
  The LUS radiographic findings will be assessed to determine a possible correlation between the radiographic findings and disease timeline, clinical symptoms such as median oxygen saturation percentage readings, the number of ER visits, and the number hospital admissions. The score from a radiographic assessment will be compared to the course of a subject's illness.

CONTACTS AND LOCATIONS:
Locations (1):
- Rocket Doctor Inc., Toronto, Ontario, Canada

REFERENCES:
- [Derived] Elmi N, Sadri Y, Myslik F, Chenkin J, Cherniak W. Self-administered at-home lung ultrasound with remote guidance in patients without clinical training. Respir Res. 2024 Mar 5;25(1):111. doi: 10.1186/s12931-024-02744-y. PMID 38443957